CLINICAL TRIAL: NCT00455429
Title: A Double-Blind, Randomized, Placebo-Controlled, Sequential Cohort Exploratory Study of the Safety and Efficacy of JNJ-26113100 in the Treatment of Adult Atopic Dermatitis That is Moderate in Severity
Brief Title: An Efficacy and Safety Study of JNJ-26113100 in the Treatment of Adult Atopic Dermatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped due to a non-clinical safety finding.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR012946; C-2006-004
Record Dates: First submitted 2007-04-01; First posted 2007-04-03 (Estimated); Results first posted 2013-07-01 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-02

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; JNJ-26113100
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- JNJ-26113100 (50 mg) once daily (Experimental)
  Interventions: Drug: JNJ-26113100 (50 mg) once daily
- JNJ-26113100 (100 mg) once daily (Experimental)
  Interventions: Drug: JNJ-26113100 (100 mg) once daily
- JNJ-26113100 (100 mg) twice daily (Experimental)
  Interventions: Drug: JNJ-26113100 (100 mg) twice daily
- JNJ-26113100 (250 mg) twice daily (Experimental)
  Interventions: Drug: JNJ-26113100 (250 mg) twice daily

INTERVENTIONS:
Drug: Placebo — Matching placebo capsules to JNJ-26113100 (50 milligram [mg]) orally once daily or 100 mg orally once daily or 100 mg orally twice daily or 250 mg orally twice daily for 6 weeks.
  Arms: Placebo
Drug: JNJ-26113100 (50 mg) once daily — JNJ-26113100 (50 mg) capsules orally once daily for 6 weeks.
  Arms: JNJ-26113100 (50 mg) once daily
Drug: JNJ-26113100 (100 mg) once daily — JNJ-26113100 (100 mg) capsules orally once daily for 6 weeks.
  Arms: JNJ-26113100 (100 mg) once daily
Drug: JNJ-26113100 (100 mg) twice daily — JNJ-26113100 (100 mg) capsules orally twice daily for 6 weeks.
  Arms: JNJ-26113100 (100 mg) twice daily
Drug: JNJ-26113100 (250 mg) twice daily — JNJ-26113100 (250 mg) capsules orally twice daily for 6 weeks.
  Arms: JNJ-26113100 (250 mg) twice daily

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of four dose regimens (pattern of giving treatment) of JNJ-26113100 in the treatment of adult Atopic Dermatitis ([AD]; skin rash, inflammation) that is moderate in severity.

DETAILED DESCRIPTION:
This study is a double-blind (neither the researchers nor the participants know what treatment the participant is receiving), randomized (study drug assigned by chance), placebo-controlled (an inactive substance; a pretend treatment [with no drug in it] that is compared in a clinical trial with a drug to test if the drug has a real effect), sequential cohort exploratory study to evaluate the safety and effectiveness of JNJ-26113100 in the treatment of adult AD that is moderate in severity, including its effect on inflammatory biomarkers (biological molecule found in blood, other body fluids, or tissues that is a sign of a normal or abnormal process, or of a condition or disease). Participants will be sequentially assigned to 50 milligram (mg) once daily, 100 mg once daily, 100 mg twice daily or 250 mg twice daily cohort and randomly assigned to receive JNJ-26113100 or matching placebo.

The total duration of the study will be approximately 8 weeks. Participants will be asked to follow-up at the end of Week 1, 2, 3, 4, 5 and 6. A study termination visit (Day 57) will be conducted at the end of Week 8. Skin biopsies from atopic dermatitis lesions will be collected during the study to assess changes in the inflammatory disease state. Participants developing flares of their disease may be treated with triamcinolone acetonide 0.1 percent ointment twice daily for up to 7 days. Efficacy will be assessed using Investigator's Global Assessment (IGA), Eczema Area and Severity Index (EASI) and Visual Analog Scale (VAS). Blood and urine samples will be collected for standard safety laboratory tests, to measure the level of drug and effect of the drug on inflammatory biomarkers. Participant's safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:-Adult participants with Atopic Dermatitis (skin rash, inflammation) involving greater than or equal to 10 percent body surface area

* Female participants must have a negative serum pregnancy test at screening
* With the exception of well-controlled asthma, allergic rhinitis and food allergies, participants must be in good general health prior to study participation with no clinically significant abnormalities as assessed by the investigator and determined by medical history, physical examination, blood chemistry, complete blood count, coagulation tests, urinalysis and electrocardiogram (ECG)
* Male subjects must consent to utilize a medically acceptable method of contraception throughout the study including the washout period and for three months after the study is completed
* Female participants of child bearing potential must consent to utilize a medically acceptable method of contraception throughout the study including the washout period and for three months after the study is completed Exclusion Criteria:-Evidence of clinically significant hepatic, reproductive, gastrointestinal, renal, hematologic, pulmonary, neurologic, respiratory (with the exception of well-controlled asthma), endocrine or cardiovascular abnormalities or psychiatric disorders
* Participants with screening alanine aminotransferase, alkaline phosphatase or direct bilirubin levels above the upper limit of normal
* Evidence of any skin condition that in the opinion of the investigator would interfere with assessment of atopic dermatitis
* Use of any investigational drugs within the previous 30 days prior to dosing or within a period of less than five times the drug's half-life, whichever is longer
* Use of any biologic within a period of 5 times its half-life

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2007-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development L.L.C Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (19):
- United States (19):
  - Huntsville, Alabama
  - Los Angeles, California
  - Sacramento, California
  - San Diego, California
  - Stanford, California
  - Vista, California
  - Jacksonville, Florida
  - Chicago, Illinois
  - Skokie, Illinois
  - Albuquerque, New Mexico
  - Rochester, New York
  - Stony Brook, New York
  - Sylvania, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - College Station, Texas
  - San Antonio, Texas
  - Seattle, Washington
  - Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching placebo capsules to JNJ-26113100 (50 milligram [mg]) orally once daily or 100 mg orally once daily or 100 mg orally twice daily for 6 weeks.
Period: Overall Study
Arm/Group | Placebo | JNJ-26113100 (50 mg) Once Daily | JNJ-26113100 (100 mg) Once Daily | JNJ-26113100 (100 mg) Twice Daily
Started | 18 | 15 | 17 | 34
Treated | 18 | 15 | 17 | 32
Completed | 16 | 10 | 16 | 20
Not Completed | 2 | 5 | 1 | 14
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 3
Not completed — Lost to Follow-up | 1 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 3
Not completed — Randomly assigned but not treated | 0 | 0 | 0 | 2
Not completed — Personal Reason | 1 | 0 | 0 | 0
Not completed — Non-compliance | 0 | 0 | 0 | 1
Not completed — Other | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | JNJ-26113100 (50 mg) Once Daily | JNJ-26113100 (100 mg) Once Daily | JNJ-26113100 (100 mg) Twice Daily | Total
Number analyzed (Participants) | 18 | 15 | 17 | 34 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (11.84) | 34.8 (14.67) | 34.6 (13.98) | 38.7 (14.50) | 36.0 (13.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 11 | 21 | 47
  Male | 8 | 10 | 6 | 13 | 37

OUTCOME MEASURES:

1. Primary Outcome: Investigator's Global Assessment (IGA) Score at Week 6
Description: Participants were reported for IGA. IGA is an overall assessment of Atopic Dermatitis (AD). IGA utilizes a 6-point scale (ranging from 0 to 5): 0=clear (noinflammatory signs of AD), 1=almost clear (just perceptible erythema, and just perceptible papulation/infiltration), 2=mild disease (mild erythema, and mild papulation/infiltration), 3=moderate disease (moderate erythema, and moderate papulation/infiltration), 4=severe disease (severe erythema, and severe papulation/infiltration) and 5=very severe disease (severe erythema, and severe papulation/infiltration with oozing/crusting).
Time Frame: Week 6
Population: Efficacy evaluable analysis set included participants who had at least 1 efficacy assessment during the dosing period. Last Observation Carried Forward (LOCF) method was used.
Measure: Number; unit: participants
Arm/Group | Placebo | JNJ-26113100 (50 mg) Once Daily | JNJ-26113100 (100 mg) Once Daily | JNJ-26113100 (100 mg) Twice Daily
Number analyzed (Participants) | 18 | 15 | 17 | 32
participants
  Clear | 1 | 1 | 1 | 2
  Almost Clear | 3 | 4 | 2 | 4
  Mild Disease | 5 | 3 | 4 | 5
  Moderate Disease | 7 | 6 | 9 | 19
  Severe Disease | 2 | 1 | 1 | 2
Statistical Analysis 1: Comparison: Placebo vs JNJ-26113100 (50 mg) Once Daily; Test type: Superiority or Other; p = 0.600, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs JNJ-26113100 (100 mg) Once Daily; Test type: Superiority or Other; p = 0.822, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs JNJ-26113100 (100 mg) Twice Daily; Test type: Superiority or Other; p = 0.656, Cochran-Mantel-Haenszel

2. Primary Outcome: Change From Baseline in Eczema Area and Severity Index (EASI) Score at Week 6
Description: EASI measures erythema (E), infiltration (I), excoriation (Ex) and lichenification (L) on a scale of 0 (none) to 3 (severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no eruption) to 6 (greater than [>] 90%-100% eruption). The total score is the sum of the four body-region scores, maximum=72, minimum=0, with higher scores reflecting greater disease severity. The total qualitative score is multiplied by the degree of involvement for each anatomic region and then multiplied by a constant and summed to yield the EASI score.
Time Frame: Baseline and Week 6
Population: Efficacy evaluable analysis set included participants who had at least 1 efficacy assessment during the dosing period. LOCF method was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | JNJ-26113100 (50 mg) Once Daily | JNJ-26113100 (100 mg) Once Daily | JNJ-26113100 (100 mg) Twice Daily
Number analyzed (Participants) | 18 | 15 | 17 | 32
units on a scale
  Baseline | 13.7 (10.93) | 12.6 (6.63) | 14.3 (9.32) | 17.2 (12.23)
  Change at Week 6 | -2.3 (5.97) | -5.5 (5.78) | -3.7 (7.18) | -4.2 (9.67)
Statistical Analysis 1: Comparison: Placebo vs JNJ-26113100 (50 mg) Once Daily; Test type: Superiority or Other; p = 0.427, Dunnett-Hsu; LS Mean difference = -3.4, 95% CI 2-sided [-9.70 to 2.90], Standard Error of Mean 2.63
Statistical Analysis 2: Comparison: Placebo vs JNJ-26113100 (100 mg) Once Daily; Test type: Superiority or Other; p = 0.922, Dunnett-Hsu; LS Mean Difference = -1.3, 95% CI 2-sided [-7.37 to 4.82], Standard Error of Mean 2.55
Statistical Analysis 3: Comparison: Placebo vs JNJ-26113100 (100 mg) Twice Daily; Test type: Superiority or Other; p = 0.919, Dunnett-Hsu; LS Mean Difference = -1.1, 95% CI 2-sided [-6.49 to 4.21], Standard Error of Mean 2.24

3. Primary Outcome: Change From Baseline in Visual Analog Scale (VAS) Score for Pruritus at Week 6
Description: VAS consists of 10 centimeter (cm) horizontal line and the words; 0 cm="No itch" on the left side of the line and the words 10 cm="Worst possible itch" on the right side of the line. Participants will be instructed to rate the severity of their pruritus within the previous 24 hours by drawing a vertical line across the 10 cm line at the point between "No itch" and "Worst possible itch" which best describes their itching during the preceding 24 hours.
Time Frame: Baseline and Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Placebo | JNJ-26113100 (50 mg) Once Daily | JNJ-26113100 (100 mg) Once Daily | JNJ-26113100 (100 mg) Twice Daily
Number analyzed (Participants) | 18 | 15 | 17 | 32
millimeter (mm)
  Baseline | 49.4 (27.94) | 47.9 (27.78) | 65.3 (18.37) | 63.4 (23.02)
  Change at Week 6 | -24.8 (32.44) | -19.9 (31.16) | -22.8 (26.66) | -20.6 (29.18)
Statistical Analysis 1: Comparison: Placebo vs JNJ-26113100 (50 mg) Once Daily; Test type: Superiority or Other; p = 0.941, Dunnett-Hsu; LS Mean difference = 3.7, 95% CI 2-sided [-15.83 to 23.18], Standard Error of Mean 8.15
Statistical Analysis 2: Comparison: Placebo vs JNJ-26113100 (100 mg) Once Daily; Test type: Superiority or Other; p = 0.196, Dunnett-Hsu; LS Mean Difference = 14.2, 95% CI 2-sided [-5.12 to 33.52], Standard Error of Mean 8.07
Statistical Analysis 3: Comparison: Placebo vs JNJ-26113100 (100 mg) Twice Daily; Test type: Superiority or Other; p = 0.096, Dunnett-Hsu; LS Mean Difference = 14.9, 95% CI 2-sided [-2.00 to 31.86], Standard Error of Mean 7.08

4. Primary Outcome: Percentage of Participants Achieving Treatment Response as "Clear" or "Almost Clear "in IGA
Description: Percentage of participants achieving treatment response (decrease) in IGA were assessed. IGA is used to assess AD through a 6-point scale (Range=0-5) where, 0=clear (no inflammatory signs of AD), 1=almost clear (just perceptible erythema & perceptible papulation/infiltration), 2=mild (mild erythema & papulation/infiltration), 3=moderate (moderate erythema & papulation/infiltration), 4=severe (severe erythema & papulation/infiltration) & 5=very severe (severe erythema & papulation/infiltration with oozing/crusting). Success is reduction of IGA to 0 or 1. Failure is reduction of IGA to >=2.
Time Frame: Baseline up to Week 6
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-26113100 (50 mg) Once Daily | JNJ-26113100 (100 mg) Once Daily | JNJ-26113100 (100 mg) Twice Daily
Number analyzed (Participants) | 18 | 15 | 17 | 32
percentage of participants
  Success | 27.8 (27.94) | 40.0 (27.78) | 17.6 (18.37) | 18.8 (23.02)
  Failure | 72.2 (32.44) | 60.0 (31.16) | 82.4 (26.66) | 81.3 (29.18)
Statistical Analysis 1: Comparison: Placebo vs JNJ-26113100 (50 mg) Once Daily; Test type: Superiority or Other; p = 0.460, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs JNJ-26113100 (100 mg) Once Daily; Test type: Superiority or Other; p = 0.479, Regression, Logistic
Statistical Analysis 3: Comparison: Placebo vs JNJ-26113100 (100 mg) Twice Daily; Test type: Superiority or Other; p = 0.462, Regression, Logistic

5. Primary Outcome: Percentage of Participants Achieving 50% Reduction in EASI Score at Week 6
Description: EASI measures erythema (E), infiltration (I), excoriation (Ex) and lichenification (L) on a scale of 0 (none) to 3 (severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no eruption) to 6 (greater than [>] 90%-100% eruption). The total score is the sum of the four body-region scores, maximum=72, minimum=0, with higher scores reflecting greater disease severity. The total qualitative score is multiplied by the degree of involvement for each anatomic region and then multiplied by a constant and summed to yield the EASI score. Success is defined as an improvement of >=50% from the baseline EASI score. An improvement of <50% is considered a failure.
Time Frame: Baseline up to Week 6
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-26113100 (50 mg) Once Daily | JNJ-26113100 (100 mg) Once Daily | JNJ-26113100 (100 mg) Twice Daily
Number analyzed (Participants) | 18 | 15 | 17 | 32
percentage of participants
  Success | 44.4 (27.94) | 60.0 (27.78) | 41.2 (18.37) | 31.3 (23.02)
  Failure | 55.6 (32.44) | 40.0 (31.16) | 58.8 (26.66) | 68.8 (29.18)
Statistical Analysis 1: Comparison: Placebo vs JNJ-26113100 (50 mg) Once Daily; Test type: Superiority or Other; p = 0.363, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs JNJ-26113100 (100 mg) Once Daily; Test type: Superiority or Other; p = 0.968, Regression, Logistic
Statistical Analysis 3: Comparison: Placebo vs JNJ-26113100 (100 mg) Twice Daily; Test type: Superiority or Other; p = 0.501, Regression, Logistic

6. Primary Outcome: Percentage of Participants Achieving Greater Than (>) or Equal to (=) 25% Reduction in EASI Score at Week 6
Description: EASI measures erythema (E), infiltration (I), excoriation (Ex) and lichenification (L) on a scale of 0 (none) to 3 (severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no eruption) to 6 (greater than [>] 90%-100% eruption). The total score is the sum of the four body-region scores, maximum=72, minimum=0, with higher scores reflecting greater disease severity. The total qualitative score is multiplied by the degree of involvement for each anatomic region and then multiplied by a constant and summed to yield the EASI score. Success is defined as an improvement of >=25% from the baseline EASI score. An improvement of <25% is considered a failure.
Time Frame: Baseline up to Week 6
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-26113100 (50 mg) Once Daily | JNJ-26113100 (100 mg) Once Daily | JNJ-26113100 (100 mg) Twice Daily
Number analyzed (Participants) | 18 | 15 | 17 | 32
percentage of participants
  Success | 55.6 (27.94) | 73.3 (27.78) | 64.7 (18.37) | 40.6 (23.02)
  Failure | 44.4 (32.44) | 26.7 (31.16) | 35.3 (26.66) | 59.4 (29.18)
Statistical Analysis 1: Comparison: Placebo vs JNJ-26113100 (50 mg) Once Daily; Test type: Superiority or Other; p = 0.333, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs JNJ-26113100 (100 mg) Once Daily; Test type: Superiority or Other; p = 0.527, Regression, Logistic
Statistical Analysis 3: Comparison: Placebo vs JNJ-26113100 (100 mg) Twice Daily; Test type: Superiority or Other; p = 0.353, Regression, Logistic

7. Primary Outcome: Percentage of Participants Achieving Greater Than (>) or Equal to (=) 75% Reduction in VAS Score for Pruritus at Week 6
Description: VAS consists of 10 centimeter (cm) horizontal line and the words; 0 cm="No itch" on the left side of the line and the words 10 cm="Worst Possible Itch" on the right side of the line. Participants will be instructed to rate the severity of their pruritus within the previous 24 hours by drawing a vertical line across the 10 cm line at the point between "No itch" and "Worst possible itch" which best describes their itching during the preceding 24 hours. Success is defined as an improvement of >=75% from the baseline VAS assessment of pruritus. An improvement of <75% is a failure.
Time Frame: Baseline up to Week 6
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-26113100 (50 mg) Once Daily | JNJ-26113100 (100 mg) Once Daily | JNJ-26113100 (100 mg) Twice Daily
Number analyzed (Participants) | 18 | 15 | 17 | 31
percentage of participants
  Success | 27.8 (27.94) | 20.0 (27.78) | 23.5 (18.37) | 12.9 (23.02)
  Failure | 72.2 (32.44) | 80.0 (31.16) | 76.5 (26.66) | 87.1 (29.18)
Statistical Analysis 1: Comparison: Placebo vs JNJ-26113100 (50 mg) Once Daily; Test type: Superiority or Other; p = 0.631, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs JNJ-26113100 (100 mg) Once Daily; Test type: Superiority or Other; p = 0.523, Regression, Logistic
Statistical Analysis 3: Comparison: Placebo vs JNJ-26113100 (100 mg) Twice Daily; Test type: Superiority or Other; p = 0.101, Regression, Logistic

8. Primary Outcome: Percentage of Participants Achieving Greater Than (>) or Equal to (=) 50% Reduction in VAS Score for Pruritus at Week 6
Description: as for outcome 7
Time Frame: Baseline up to Week 6
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-26113100 (50 mg) Once Daily | JNJ-26113100 (100 mg) Once Daily | JNJ-26113100 (100 mg) Twice Daily
Number analyzed (Participants) | 18 | 15 | 17 | 31
percentage of participants
  Success | 50.0 (27.94) | 60.0 (27.78) | 41.2 (18.37) | 38.7 (23.02)
  Faliure | 50.0 (32.44) | 40.0 (31.16) | 58.8 (26.66) | 61.3 (29.18)
Statistical Analysis 1: Comparison: Placebo vs JNJ-26113100 (50 mg) Once Daily; Test type: Superiority or Other; p = 0.429, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs JNJ-26113100 (100 mg) Once Daily; Test type: Superiority or Other; p = 0.206, Regression, Logistic
Statistical Analysis 3: Comparison: Placebo vs JNJ-26113100 (100 mg) Twice Daily; Test type: Superiority or Other; p = 0.107, Regression, Logistic

9. Primary Outcome: Percentage of Participants Achieving Greater Than (>) or Equal to (=) 25% Reduction in VAS Score for Pruritus at Week 6
Description: as for outcome 7
Time Frame: Baseline up to Week 6
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-26113100 (50 mg) Once Daily | JNJ-26113100 (100 mg) Once Daily | JNJ-26113100 (100 mg) Twice Daily
Number analyzed (Participants) | 18 | 15 | 17 | 31
percentage of participants
  Success | 55.6 (27.94) | 73.3 (27.78) | 41.2 (18.37) | 58.1 (23.02)
  Failure | 44.4 (32.44) | 26.7 (31.16) | 58.8 (26.66) | 41.9 (29.18)
Statistical Analysis 1: Comparison: Placebo vs JNJ-26113100 (50 mg) Once Daily; Test type: Superiority or Other; p = 0.097, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs JNJ-26113100 (100 mg) Once Daily; Test type: Superiority or Other; p = 0.077, Regression, Logistic
Statistical Analysis 3: Comparison: Placebo vs JNJ-26113100 (100 mg) Twice Daily; Test type: Superiority or Other; p = 0.489, Regression, Logistic

10. Primary Outcome: Percentage of Participants Who Had at Least 1 Flare
Description: Percentage of participants who had at Least 1 Flare while on treatment was assessed. A flare was considered to be present if the following criteria were met: 1) IGA was greater than or equal to 2, if IGA on most recent previous assessment was 0; 2) IGA had increased by at least 1 point, if IGA on most recent previous assessment was 1 or more.
Time Frame: Baseline up to Week 6
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-26113100 (50 mg) Once Daily | JNJ-26113100 (100 mg) Once Daily | JNJ-26113100 (100 mg) Twice Daily
Number analyzed (Participants) | 18 | 15 | 17 | 32
percentage of participants
  YES | 50.0 (27.94) | 60.0 (27.78) | 35.3 (18.37) | 34.4 (23.02)
  NO | 50.0 (32.44) | 40.0 (31.16) | 64.7 (26.66) | 65.6 (29.18)
Statistical Analysis 1: Comparison: Placebo vs JNJ-26113100 (50 mg) Once Daily; Test type: Superiority or Other; p = 0.566, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs JNJ-26113100 (100 mg) Once Daily; Test type: Superiority or Other; p = 0.382, Regression, Logistic
Statistical Analysis 3: Comparison: Placebo vs JNJ-26113100 (100 mg) Twice Daily; Test type: Superiority or Other; p = 0.282, Regression, Logistic

11. Primary Outcome: Number of Flare Occurrences Per Participant
Description: A flare was considered to be present if the following criteria were met: 1) IGA was greater than or equal to 2, if IGA on most recent previous assessment was 0 or 2) IGA had increased by at least 1 point, if IGA on most recent previous assessment was 1 or more.
Time Frame: Baseline up to Week 6
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | JNJ-26113100 (50 mg) Once Daily | JNJ-26113100 (100 mg) Once Daily | JNJ-26113100 (100 mg) Twice Daily
Number analyzed (Participants) | 18 | 15 | 17 | 32
participants
  0 flare | 9 (27.94) | 6 (27.78) | 11 (18.37) | 21 (23.02)
  1 flare | 6 (32.44) | 3 (31.16) | 4 (26.66) | 9 (29.18)
  2 flares | 3 | 5 | 2 | 1
  3 flares | 0 | 1 | 0 | 1
Statistical Analysis 1: Comparison: Placebo vs JNJ-26113100 (50 mg) Once Daily; Test type: Superiority or Other; p = 0.206, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs JNJ-26113100 (100 mg) Once Daily; Test type: Superiority or Other; p = 0.433, Regression, Logistic
Statistical Analysis 3: Comparison: Placebo vs JNJ-26113100 (100 mg) Twice Daily; Test type: Superiority or Other; p = 0.290, Regression, Logistic

12. Primary Outcome: Percentage of Participants Who Had at Least 1 Worsening AD Event
Description: Percentage of Participants who had at least 1 Worsening AD Event That did not Meet Flare Criteria were assessed. Worsening of AD that did not meet flare criteria was documented. Flare was considered to be present if either of the following criteria were met: 1) IGA was=2, if IGA on most recent previous assessment was 0; 2) IGA had increased by at least 1 point, if IGA on most recent previous assessment was 1 or more.
Time Frame: Baseline up to Week 6
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-26113100 (50 mg) Once Daily | JNJ-26113100 (100 mg) Once Daily | JNJ-26113100 (100 mg) Twice Daily
Number analyzed (Participants) | 18 | 15 | 17 | 32
percentage of participants
  YES | 11.1 (27.94) | 20.0 (27.78) | 11.8 (18.37) | 21.9 (23.02)
  NO | 88.9 (32.44) | 80.0 (31.16) | 88.2 (26.66) | 78.1 (29.18)
Statistical Analysis 1: Comparison: Placebo vs JNJ-26113100 (50 mg) Once Daily; Test type: Superiority or Other; p = 0.484, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs JNJ-26113100 (100 mg) Once Daily; Test type: Superiority or Other; p = 0.952, Regression, Logistic
Statistical Analysis 3: Comparison: Placebo vs JNJ-26113100 (100 mg) Twice Daily; Test type: Superiority or Other; p = 0.350, Regression, Logistic

13. Secondary Outcome: Plasma Concentration of JNJ-26113100
Description: Blood samples for pharmacokinetic (PK) analysis were collected before dosing and at 0.25 to 3 hours after dosing at randomization (Day 1) and Week 3 visit and at 0.25 to 3 hours, 4 to 6 hours, and 7 to 12 hours after dosing at Week 6.
Time Frame: Before dosing on Day 1, Week 3, Week 6; after dosing at 0.25 to 3 hours on Day 1, Week 3, Week 6; after dosing at 4 to 6 hours and 7 to 12 hours on Week 6
Population: Intent-to-treat (ITT) analysis set included all participants who were randomly assigned to treatment groups and received at least 1 dose of study drug. LOCF method was used.
Measure: Mean (Standard Deviation); unit: nanogram (ng)/milli litre (mL)
Arm/Group | JNJ-26113100 (50 mg) Once Daily | JNJ-26113100 (100 mg) Once Daily | JNJ-26113100 (100 mg) Twice Daily
Number analyzed (Participants) | 15 | 17 | 30
nanogram (ng)/milli litre (mL)
  Predose (Day 1) | NA (NA) — For all participants the plasma concentration was below quantifiable limit (BQL [1 ng/ml]). Lower limit of quantification = 1.0 ng/mL. | NA (NA) — For all participants the plasma concentration was below quantifiable limit (BQL [1 ng/ml]). Lower limit of quantification = 1.0 ng/mL. | 1.07 (NA) — Only one participant had plasma concentration above the below quantifiable limit (BQL [1ng/ml]). Lower limit of quantification = 1.0 ng/mL.
  Postdose (0.25 - 3 h, Day 1) | 228 (249) | 979 (1089) | 787 (1262)
  Predose (Week 3) | 43.0 (28.2) | 324 (328) | 665 (683)
  Postdose (0.25 - 3 h, Week 3) | 195 (402) | 1050 (962) | 1542 (1406)
  Predose (Week 6) | 112 (103) | 346 (472) | 965 (732)
  Postdose (0.25 - 3 h, Week 6) | 285 (261) | 1420 (1734) | 1475 (1486)
  Postdose (4 - 6 h, Week 6) | 630 (318) | 1889 (976) | 1728 (867)
  Postdose (7 -12 h, Week 6) | 417 (196) | 1182 (676) | 1305 (703)

ADVERSE EVENTS:
Time Frame: From signing of informed consent until the study termination visit (Day 57)
Arm/Group | Placebo | JNJ-26113100 (50 mg) Once Daily | JNJ-26113100 (100 mg) Once Daily | JNJ-26113100 (100 mg) Twice Daily
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/15 | 0/17 | 0/32
Other Adverse Events (participants affected / at risk) | 12/18 | 10/15 | 14/17 | 31/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=18) | JNJ-26113100 (50 mg) Once Daily (N=15) | JNJ-26113100 (100 mg) Once Daily (N=17) | JNJ-26113100 (100 mg) Twice Daily (N=32)
Nasopharyngitis (Infections and infestations) | 2 | 0 | 2 | 5
Urinary tract infection (Infections and infestations) | 0 | 0 | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 2 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 1
Abscess (Infections and infestations) | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 | 3 | 3 | 7
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Tooth impacted (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Anal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 1 | 2 | 3
Urine albumin/creatinine ratio increased (Investigations) | 1 | 0 | 1 | 4
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 2 | 1 | 2 | 3
Hypoesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 2 | 1
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0
Edema peripheral (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Foreign body trauma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Participants were not enrolled into JNJ-26113100(250 mg) twice daily dose because the study was stopped during 100mg twice daily dose due to preclinical finding of retinal atrophy in high dose group(150 mg/kg) of 6-month, albino rat toxicology study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days